CLINICAL TRIAL: NCT02597699
Title: Use of Ultiva ® Associated With Xylocaine ® in the Procedures of Feticide: A Phase III Randomized Trial
Brief Title: Use of Ultiva ® Associated With Xylocaine ® in the Procedures of Feticide
Acronym: FOETIVA2
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital, Montpellier (Other)
Collaborators: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 94602; 2015-002856-28 (EudraCT Number)
Record Dates: First submitted 2015-10-27; First posted 2015-11-05 (Estimated); Last update posted 2025-10-03 (Actual); Status verified 2025-09

CONDITIONS: Termination of Pregnancy; Feticide
Keywords: Termination of pregnancy; Feticide; Fetal pain; Remifentanil Ultiva®; Fetal asystole; Fetopathologic analysis
MeSH Terms: interventions — Remifentanil; Sufentanil

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm 1: Sufentanil + Lidocaïne (Active Comparator): For patients randomized to arm 1, as in the current practice, we will inject Sufentanil intra-cordially at the dose of 1.5 μg / kg of the estimated fetal weight, then the Lidocaïne 1% bolus of 10 ml (10 mg / ml).
  If 2 minutes after the start of the injection of Lidocaïne, there is no obtaining of fetal asystole, we will inject 100mg of Lidocaïne 1% in bolus of 10 ml. In the event of failure of the procedure, we will inject 10ml of KCL 10% intra-cordial if the cord is always accessible, if not intra-cardiac.
  Interventions: Drug: Sufentanil + Lidocaïne
- Arm 2: Remifentanil + Lidocaïne (Experimental): For patients randomized to arm 2, we will inject 30 μg of intravenous Remifentanil (Ultiva®) followed by Xylocaine 1% in a 10 ml bolus (10 mg / ml).
  If 2 minutes after the start of the injection of Lidocaïne, there is no obtaining of asystole, we will inject 100 mg of Lidocaïne 1% in bolus of 10 ml. In case of failure of the procedure, we will inject 10 ml of KCL 10% intra-cordial if the cord is still accessible, if not intra-cardiac.
  Interventions: Drug: Remifentanil + Lidocaïne

INTERVENTIONS:
Drug: Remifentanil + Lidocaïne
  Other Names: Ultiva® + Xylocaïne®
  Arms: Arm 2: Remifentanil + Lidocaïne
Drug: Sufentanil + Lidocaïne
  Other Names: Sufentanil + Xylocaïne®
  Arms: Arm 1: Sufentanil + Lidocaïne

SUMMARY:
The feticide is a legal and ethical obligation during a termination of pregnancy after 22 weeks' gestation. This method raise concerns about the fetal pain, maternal complications and the fetopathologic analysis. There are few studies on the subject. Investigators want to evaluate a drug in order to facilitate this method technically and emotionally challenging. They want to achieve a quick fetal asystole, a fetal analgesia, a maternal security and a optimal fetopathologic analysis. A drug, remifentanil Ultiva®, seems could meet its properties, it is a powerful morphine. A phase 2 clinical trial has assessed the feasibility, efficacy and safety of Ultiva®. They had not been able to prove bradycardia or lethal effect of Ultiva injected alone but the feasibility and safety were good.

Investigators want to set up a randomized clinical trial with 2 arms : Ultiva® and lidocaine versus sufentanil and lidocaine (standard protocol), it is a bicentric study. The primary outcome is the interval between the vascular injection of lidocaine and fetal asystole. The secondary outcomes are the success rate of method, the number of puncture of the umbilical cord, the maternal side effects and the quality of fetopathologic analysis.

The previous observational study showed a median interval of 2,3 minutes and a success rate of 55% (lower interval to 2 minutes). From the results they calculate a necessary inclusions to 66 patients.

They believe that the bradycardia property of Ultiva® allow a potentiation of the efficacy of lidocaine. If the results are satisfactory, the use of Ultiva® can be generalized to other fetal medicine team.

DETAILED DESCRIPTION:
The intervention will take place, as in the framework of usual care, obstetric block after achievement of maternal locoregional anesthesia peri-rachianesthesia, skin disinfection and sterile field. The gesture will be performed by an experienced obstetrician under ultrasound guidance. Anesthetist-resuscitator is present in the obstetric block. Peri-rachianesthesia is performed by the initial injection of 2.5mg of hyperbaric bupivacaine associated with 5 gamma of Sufentanil and 0.5ml of physiological saline.

Inclusion in one of two arms is defined after randomization in single blind:

Arm 1 (Sufentanil + Lidocaïne) or Arm 2 (Ultiva® + Lidocaïne) For patients randomized in the arm 1, we will realize the reference protocol, as in the current practice, by injecting Sufentanil intra-cordally at the posology of 1,5 μg / kg of estimated fetal weight, then Lidocaïne 1% in bolus of 10 ml (10 mg / ml).

If 2 minutes after the start of the injection of Lidocaïne, there is no obtaining of fetal asystole, we will inject 100 mg of Lidocaïne 1% into a 10 ml bolus. In case of failure of the procedure, we will inject 10ml of KCL 10% intra-cordial if the cord is still accessible, if not intra-cardiac.

For patients randomized to arm 2, we will intracenally inject Ultiva® 30 μg and Lidocaïne 1% into 10 ml bolus (10 mg / ml).

If 2 minutes after the start of the injection of Lidocaïne, there is no obtaining of asystole, we will inject 100 mg of Lidocaïne 1% in 10 ml bolus. In case of failure of the procedure, we will inject 10 ml of KCL 10% intra-cordally if the cord is still accessible, if not intra-cardiac.

ELIGIBILITY:
Inclusion Criteria:

1. Age > = 18 years
2. Patient having received an authorization of medical termination of pregnancy beyond 22 weeks of amenorrhea by the Multidisciplinary Centers of Prenatal Diagnosis of Montpellier or Nimes
3. Patient member or beneficiary of a national insurance scheme
4. Patient capable of understanding the nature, the purpose and the methodology of the trial
5. Patient having given an informed consent signed before the inclusion in the trial

Exclusion Criteria:

1. Patient presenting a selective or total feticide in the cases of multiple pregnancies (the first preferential way in these cases is intracardiac, moreover the act risks to be complicated by the active movements of the other foetus)
2. Major Patient protected by the law (guardianship, curators, or under protection of justice)
3. Patient deprived of freedom by court or administrative order

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2015-12-18 (Actual); Primary Completion 2019-03-07 (Actual); Study Completion 2019-05-06 (Actual)

PRIMARY OUTCOMES:
The deadline of obtaining the asystole | up to 5 minutes
  The deadline of obtaining the asystole after the beginning of the injection of the ULTIVA associated with Xylocaine versus the reference protocol Sufentanil and Xylocaine

SECONDARY OUTCOMES:
The success rate of the procedure of foeticide | within 2 minutes after injection of Lidocaïne and persistent during at least 1 minute
  Fetal asystole after injection of Lidocaïne and persisted for at least 1 minute. Fetal asystole should be confirmed by the birth of a non-living fetus during delivery.
The number of new punction(s) of the cordon | 1 day
  The number of new puncture(s) of the cord, after injection of the necessary lethal agent before persistent fetal heart failure.
Number of side effects | 1 day
  Number of serious side effects in patients
The quality of tissues (the fetopathologic analysis) | 1 day
  The presence of abnormal tissue(s) or cell(s) may alter the quality of the fetopathological examination. Macroscopic examination of tissues will be performed blind of the procedure used for feticide, the only anomaly described so far in feticides is the presence of whitish deposits when using KCL.

CONTACTS AND LOCATIONS:
Overall Officials: Romy RR RAYSSIGUIER, MD, Principal Investigator — Montpellier University Hospital
Locations (2):
- France (2):
  - Hôpital Arnaud de Villeneuve, Montpellier
  - Nîmes University Hospital, Nîmes

REFERENCES:
- [Result] Rayssiguier R, Fuchs F, Mousty E, Morau E, Hlioua T, Wells C, Musizzano Y, Nagot N, Graf C, Legoux C, Boulot P, Dumont C. Use of Remifentanil Associated with Lidocaine for Feticides in Late Terminations of Pregnancy: A Randomized Clinical Trial. Fetal Diagn Ther. 2021;48(11-12):812-818. doi: 10.1159/000520448. Epub 2021 Nov 22. PMID 34808620